CLINICAL TRIAL: NCT05251246
Title: Recovery Optimisation in Emergency Medicine Addressing Stress Adaptation Techniques
Brief Title: Impact of Stress and Sleep Management on Emergency Professionals
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL21_0774; 2021-A02218-33 (Other: ID-RCB)
Record Dates: First submitted 2021-11-30; First posted 2022-02-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: sleep deprivation; recovery management program; Stress, Psychological; Stress, Physiological; Emergency Service; Hospital; nurses; physicians
MeSH Terms: conditions — Sleep Deprivation; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Without recovery management program (No Intervention)
- Trained in the recovery management program (Experimental): Half of the included volunteered participants are randomized in the intervention group
  Interventions: Behavioral: recovery management program

INTERVENTIONS:
Behavioral: recovery management program — The recovery management program consists in training the nurses and physicians during a 15-day training course to optimize their recovery abilities : sleep management according to the schedules by anticipation and recovery, and stress management through cardio-feedback techniques (cardiac coherence) also called controlled breathing techniques and mental imagery.
  Arms: Trained in the recovery management program

SUMMARY:
The investigators hypothesize that a recovery management program could have an impact on emergency nurses and physicians by improving their sleep and reducing their psychological and physiological responses when dealing with stressful situations during their professional practice. The REST study consists in developing a recovery management program for emergency professionals. The following strategies would be proposed :

* sleep management according to their schedules by anticipation and recovery,
* stress management through cardio-feedback techniques (cardiac coherence) also called controlled breathing techniques and mental imagery.

The objectives are to evaluate the impact of this program on the physiological and psychological stress of the emergency professionals during their professional activity, as well as on their sleep. To do so, their respiratory and heart rates, as well as their activity and resting times will be recorded continuously for one week. At the end of each shift, the emergency professionals will report and evaluate the 3 most stressful events.

ELIGIBILITY:
Inclusion Criteria:

* Nurses or physicians
* In current position for at least one year
* Full time or minimum three shifts per week
* Location: Emergency Department of the Edouard Herriot Hospital or the South Lyon Hospital
* Free and informed consent

Exclusion Criteria:

* Caregivers on leave during the enrollment period
* Pregnant, parturient or breastfeeding caregivers
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the recovery capacity for self-reported stressful events after the recovery management program | 30 minutes post-stressful events
  During the 30 minutes following self-reported stressful events, the physiological responses to stress (heart rate) are compared between the trained and non-trained emergency professionals.

SECONDARY OUTCOMES:
Evaluation of the perceived stress of the emergency professionals across one week of shift work before and after implementation of the recovery management program. | 2 days (Day22 & Day51)
  After each monitored week of shift work, the overall perceived stress is collected once using the Perceived Stress Scale (PSS ranging from 0 minimum to 42 maximum).
Evaluation of the perceived stress of the emergency professionals during the shift work before and after implementation of the recovery management program | 6 days (each shift between Day 15 - Day 21 & Day 44-51)
  Before (baseline) and after each shift, the perceived stress during the experienced shift is collected every time using the Visual Analogue Scale VAS for stress intensity (VAS-Stress ranging from 0 minimum to 10 maximum).
Evaluation of the psychological markers of stress for self-reported stressful events before and after implementation of the recovery management program. | 6 days (between Day 15- Day 21 & Day 44-51))
  After the shift following self-reported stressful events, the psychological markers of stress are evaluated using the visual analogue scale (VAS-event ranging from 0 minimum to 10 maximum) to indicate the intensity of each event.
Comparison of the sleep time and latency of sleep times before and after implementation of the recovery management program. | 7 days (Day 15-Day 21)
  Sleep time and latency of sleep are recorded by actimetry.
Evaluation of the subjective perception of somnolence before and after implementation of the recovery management program. | 6 days (each shift between Day 15- Day 21 & Day 44-51)
  During the week of shift observation, before and after the working time, the subjective perception of somnolence is measured using the Karolinska scale (KSS ranging from 0 minimum to 9 maximum) to evaluate the impact of the recovery management program
Evaluation of mental fatigue before and after implementation of the recovery management program | 6 days (each shift between Day 15- Day 21 & Day 44-51)
  During the week of shift observation, after work time, the mental fatigue is measured using a Visual Analogue Scale (VAS ranging from 0 minimum to 10 maximum) to evaluate the impact of the recovery management program.
Evaluation of the overall sleepiness before and after implementation of the recovery management program | 2 days (Day 22 & Day 51)
  After each monitored week of shift work, the overall sleepiness is measured using the Epworth Sleepiness Scale (ESS ranging from 0 minimum to 24 maximum) to evaluate the impact of the recovery management program
Evaluation of the sleep quality before and after implementation of the recovery management program | 2 days (Day 22 & Day 51)
  After each monitored week of shift work, the overall sleep quality is measured using the Insomnia Severity Index (ISI ranging from 0 minimum to 28 maximum) to evaluate the impact of the recovery management program.
Evaluation of bedtime arousal before and after implementation of the recovery management program | 2 days (Day 22 & Day 51)
  After each monitored week of shift work the sleep quality is measured using the score on the Pre-Sleep Arousal QScale (PSAS ranging from 16 minimum to 80 maximum) to evaluate the impact of the recovery management program.
Evaluation of the evolution of the perceived quality of sleep before and after implementation of the recovery management program. | 1 day (Day 51)
  At the end of the study, the evolution of the perceived quality of sleep is measured using the Leeds questionnaire (LSEQ including VAS from 1 to 10) to evaluate the impact of the recovery management program.
Evaluation of the job satisfaction before and after implementation of the recovery management program | 2 days (Day 22 & Day 51)
  Before and after implementation of the recovery, the job satisfaction is measured using a visual analogue scale for the effort-reward imbalance marker (ranging from 0 minimum to 10 maximum) to evaluate the impact of the recovery management program.
Evaluation of the reported adverse events before and after implementation of the recovery management program | Day 15- Day 21 & Day 44-51
  Before and after implementation of the recovery, the occurrence of adverse events is measured based on the records.

CONTACTS AND LOCATIONS:
Overall Officials: Marion DOUPLAT, MD, Principal Investigator — Hospices Civils de Lyon; Stéphanie MAZZA, Prof, Study Director — Laboratoire RESHAPE, Université Lyon 1
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No